CLINICAL TRIAL: NCT02619825
Title: Non-Invasive Evaluation of Myocardial Stiffness by Elastography Pediatric Cardiology Under
Brief Title: Non-Invasive Evaluation of Myocardial Stiffness by Elastography in Pediatric Cardiology (Elasto-Pédiatrie)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-03
Record Dates: First submitted 2015-10-23; First posted 2015-12-02 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy
Keywords: Child
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic | interventions — Ultrasonography; Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 "healthy volunteers (Other): Echography and Elastography To determine physiological standards across age classes of myocardial stiffness estimated by Elastography in ultrafast (estimated right ventricular stiffness [VD] and left ventricular [LV]). This will be done in groups of children without heart condition, age group (10 children per group, four age groups [0-1mois, 1 month-1 year 1 year-5 years, 5 years-15years]).
  Interventions: Device: Echography; Device: Elastography
- Group 2 Patients CMH primitive (Other): Echography and Elastography To evaluate myocardial stiffness Elastography (RV and LV) on different groups of children (same age group) with Hypertrophic Cardiomyopathy (HCM) non obstructive primitive and examine correlations with the conventional parameters of systolic and diastolic function of both ventricles and with myocardial strain values.
  Interventions: Device: Echography; Device: Elastography
- Group 3 Patients primitive CMD: (Other): Echography and Elastography To evaluate myocardial stiffness Elastography (RV and LV) on different groups of children (same age group) with Dilated Cardiomyopathy primitive and examine correlations with the conventional parameters of systolic and diastolic function of both ventricles and with myocardial strain values.
  Interventions: Device: Echography; Device: Elastography

INTERVENTIONS:
Device: Echography — cardiac ultrasound, in two stages, with an estimate of the stiffness of the myocardium ShearWave Elastography (Aixplorer®) and measurement of all echocardiographic parameters estimated in children with a clinical ultrasound Machine
Device: Elastography — cardiac ultrasound, in two stages, with an estimate of the stiffness of the myocardium ShearWave Elastography (Aixplorer®) and

SUMMARY:
First, investigators must determine the physiological standards across age classes of myocardial stiffness estimated by Elastography in ultrafast (estimated right ventricular stiffness [VD] and left ventricular [LV]). This will be done in groups of children without heart condition, age group (10 children per group, four age groups [0-1mois, 1 month-1 year 1 year-5 years, 5 years-15years]).

Secondly, investigators will evaluate myocardial stiffness Elastography (RV and LV) on different groups of children (same age group) with cardiomyopathy and examine correlations with the conventional parameters of systolic and diastolic function of both ventricles and with myocardial strain values. The total population of the study will be 120 children (40 healthy, 80 patients).

DETAILED DESCRIPTION:
Monocenter Prospective, open-label, non-randomized. All patients included in the study have a specific consultation built around a clinical examination and echocardiography, in two stages, with estimates of the stiffness of the myocardium ShearWave Elastography (Aixplorer®) and measures of all echocardiographic parameters estimated in children with a clinical ultrasound machine (Philips and General Electric).

Following this consultation, clinic and electrocardiographic monitoring period will be observed for 30 minutes, to ensure the safety of our procedure.

Required subjects: 40 healthy volunteers + 80 = 120 persons

ELIGIBILITY:
Inclusion Criteria:

Group 1. Healthy Age criteria met by group [0-1mois, 1 month-1 year 1 year-5 years, 5 years-15years]

* consultation for heart murmur
* Recipient of a social protection scheme or entitled (excluding AME)
* Signed informed consent by the holders of parental authority

Group 2. Patients MHC nonobstructive:

* Age criteria met by group [1 month-1 year 1 year-5 years]
* Diagnostic criteria of non-obstructive HCM validated by the medical team of pediatric cardiology center (Necker)
* Recipient of a social protection scheme or entitled (excluding AME)
* Signed informed consent by the holders of parental authority

Group 3. Patients primitive CMD:

* Age criteria met by group [1 month-1 year 1 year-5 years]
* Diagnostic criteria of primary CMD validated by the medical team of pediatric cardiology center (Necker)
* Recipient of a social protection scheme or entitled (excluding AME)
* Signed informed consent

Exclusion Criteria:

Group 1. Healthy Patients:

* Age> 15 years
* Heart and Systemic Pathology identified
* metabolic and tissue pathology.
* known genetic pathology may have cardiac involvement.
* No echogenicity,
* Allergy echocardiography gel.

Group 2. Group CMH primitive Patients

* No echogenicity,,
* Allergy echocardiography gel.
* Arrhythmia.
* Pacemaker or defibrillator

Group 3. Patients primitive CMD:

* No echogenicity,,
* Allergy echocardiography gel.
* Arrhythmia.
* Pacemaker or defibrillator

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Myocardial diastolic stiffness UltrafastEcho (kPa) | through study completion, an average of 1 year
  Normal values and intra-observer variability and inter-observer variability to demonstrate that the Aixplorer® myocardial elastography provides a reproducible assessment of myocardial stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier VILLEMAIN, MD, Study Chair — LAngevin Institute
Locations (1):
- Chu Necker, Paris, France